CLINICAL TRIAL: NCT00139074
Title: Phase IV Study to Investigate if Valproate Add-on Therapy is Superior to Quetiapine Monotherapy in Acutely Manic Patients
Brief Title: Seroquel in Acute Mania: Study to Investigate if Valproate Add-On Therapy is Superior to Quetiapine Monotherapy in Acutely Manic Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: terminated due to very low recruitment rate (27 June 2006)
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D1449L00010
Record Dates: First submitted 2005-08-29; First posted 2005-08-31 (Estimated); Last update posted 2013-01-28 (Estimated); Status verified 2013-01

CONDITIONS: Bipolar Disorder
Keywords: Bipolar I Disorder (DSM-IV 296.01, DSM-IV 296.4, DSM-IV 296.61)
MeSH Terms: conditions — Bipolar Disorder | interventions — Quetiapine Fumarate; Valproic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): quetiapine fumarate monotherapy
  Interventions: Drug: Quetiapine fumarate
- 2 (Experimental): Quetiapine + sodium valproate
  Interventions: Drug: Quetiapine fumarate; Drug: sodium valproate

INTERVENTIONS:
Drug: Quetiapine fumarate — oral variable dose
  Other Names: Seroquel
Drug: sodium valproate — oral
  Arms: 2

SUMMARY:
The primary purpose is to investigate whether the addition of sodium valproate will be superior to treatment with quetiapine (Seroquel) given as monotherapy for an additional 14 days in non-responding patients after a 14 day initial treatment period with quetiapine.

PLEASE NOTE: Seroquel SR and Seroquel XR refer to the same formulation. The SR designation was changed to XR after consultation with FDA.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from a manic or mixed episode.

Exclusion Criteria:

* Patients who have not provided personal informed consent,
* Known intolerance, hypersensitivity or lack of antimanic response to sodium valproate or quetiapine fumarate,
* Involuntary admittance/detainment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2005-07; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
The number of responders in the two treatment groups (quetiapine + sodium valproate placebo/quetiapine + sodium valproate) | after 2 weeks treatment

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Rasmus Wenzer Licht, Principal Investigator — AstraZeneca; AstraZeneca Seroquel Medical Science Director, MD, Study Director — AstraZeneca
Locations (7):
- Denmark (7):
  - Research Site, Copenhagen
  - Research Site, Esbjerg
  - Research Site, Frederikssund
  - Research Site, Haderslev
  - Research Site, Hellerup
  - Research Site, Kolding
  - Researcg Site, Svendborg